CLINICAL TRIAL: NCT01002573
Title: A Multicenter, Randomized, Open-Label, Parallel, Active-Comparator Trial to Determine the Efficacy, Safety, and Pharmacokinetics of Ibuprofen Injection in Pediatric Patients
Brief Title: Safety, Efficacy, and Pharmacokinetic Study of Intravenous Ibuprofen in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPI-CL-012
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Fever
Keywords: Pediatric; Fever
MeSH Terms: conditions — Fever | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ibuprofen (Experimental): Ibuprofen, 10 mg/kg
  Interventions: Drug: ibuprofen
- Acetaminophen (Active Comparator): Acetaminophen, 10mg/kg
  Interventions: Drug: acetaminophen

INTERVENTIONS:
Drug: ibuprofen — Ibuprofen, 10 mg/kg
  Arms: ibuprofen
Drug: acetaminophen — Acetaminophen, 10mg/kg
  Other Names: APAP (acetaminophen); paracetamol
  Arms: Acetaminophen

SUMMARY:
The primary objective of the study is to determine the superiority of a single dose of intravenous ibuprofen compared to acetaminophen for the treatment of fever during the first two hours of treatment.

DETAILED DESCRIPTION:
The primary objective of the study is to determine the superiority of a single dose of intravenous ibuprofen compared to acetaminophen for the treatment of fever as measured by the area under the change in temperature versus time curve during the first 2 hours of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Have written informed consent provided by legal parent, guardian, or authorized agent prior to participation in the study or study-only related procedures.
2. Be between birth (28 weeks to < 40 weeks gestational age) to ≤ 16 years of age.
3. Have new (less than 7 days) onset of fever, documented by temperature greater than or equal to 101.0 ºF (38.3 ºC).

Exclusion Criteria:

1. Have inadequate intravenous access.
2. Have received antipyretic drug therapy within 2 hours before dosing.
3. Have any history of allergy or hypersensitivity to NSAIDs or aspirin.
4. Have received another investigational drug within the past 30 days.
5. Be otherwise unsuitable for the study, in the opinion of the Investigator.
6. Have a fever due to hyperthermia.
7. Pregnant or nursing.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2010-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Art Wheeler, M.D., Study Director — Cumberland Pharmaceuticals, Inc.
Locations (17):
- United States (17):
  - Maricopa Medical Center, Phoenix, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital of Orange County, Orange, California
  - Howard University, Washington D.C., District of Columbia
  - Jackson Memorial Hospital (U. Miami), Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Joseph M. Still Burn Center, Augusta, Georgia
  - Kosair Children's Hospital, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Children's Hospital of Michigan, Detroit, Michigan
  - Staten Island University Hospital, Staten Island, New York
  - The Children's Hospital at Saint Francis, Tulsa, Oklahoma
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - Children's Memorial Hermann Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Khalil SN, Hahn BJ, Chumpitazi CE, Rock AD, Kaelin BA, Macias CG. A multicenter, randomized, open-label, active-comparator trial to determine the efficacy, safety, and pharmacokinetics of intravenous ibuprofen for treatment of fever in hospitalized pediatric patients. BMC Pediatr. 2017 Feb 1;17(1):42. doi: 10.1186/s12887-017-0795-y. PMID 28143430

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ibuprofen | Acetaminophen
Started | 58 | 60
Completed | 47 | 53
Not Completed | 11 | 7
Not completed — Subject did not receive at least 1 dose | 11 | 7

BASELINE CHARACTERISTICS:
Population: All Treated Subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen | Acetaminophen | Total
Number analyzed (Participants) | 47 | 53 | 100
Age, Customized [Number; unit: participants]
  6 months to 2 years | 6 | 14 | 20
  2 years to 6 years | 13 | 14 | 27
  6 years to 16 years | 28 | 25 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 27 | 47
  Male | 27 | 26 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 24 | 53
  Not Hispanic or Latino | 18 | 29 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 42 | 42 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Fever Reduction
Description: Treatment of fever as measured by the area under the change in temperature versus time curve during the first two hours of treatment (AUC0-2)
Time Frame: 0 to 2 hours post-dose
Population: Some participants data was not included in the analysis due to having too few/insufficient data
Measure: Mean (Standard Deviation); unit: degree Celsius*Time
Arm/Group | Ibuprofen | Acetaminophen
Number analyzed (Participants) | 46 | 50
degree Celsius*Time | -1.5 (1.11) | -0.9 (0.89)

2. Secondary Outcome: Change From Baseline in Temperature After the First 30 Minutes of Treatment
Description: Change in temperature in patients receiving intravenous ibuprofen and acetaminophen (APAP) after the first 30 minutes of treatment.
Time Frame: 30 minutes following treatment
Population: Some participants data was not included in the analysis due to having too few/insufficient data
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Ibuprofen | Acetaminophen
Number analyzed (Participants) | 45 | 53
Celsius | -0.5 (0.50) | -0.3 (0.49)

3. Secondary Outcome: Change From Baseline in Temperature After the First 60 Minutes of Treatment
Description: Change in temperature in patients receiving intravenous ibuprofen and APAP after the first 60 minutes of treatment.
Time Frame: 60 minutes following treatment
Population: Some participants data was not included in the analysis due to having too few/insufficient data
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Ibuprofen | Acetaminophen
Number analyzed (Participants) | 45 | 53
Celsius | -0.9 (0.69) | -0.5 (0.50)

4. Secondary Outcome: Change in Temperature
Description: Change in temperature in patients receiving intravenous ibuprofen and APAP after the first 4 hours of treatment.
Time Frame: 4 hours following treatment
Population: Some participants data was not included in the analysis due to having too few/insufficient data
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Ibuprofen | Acetaminophen
Number analyzed (Participants) | 43 | 37
Celsius | -1.5 (0.92) | -0.9 (0.92)

5. Secondary Outcome: Change From Baseline in Temperature After the First Four Hours of Treatment
Description: Change in temperature during the first 4 hours of treatment by assessing the area under the change in temperature versus time curve during the first four hours of treatment (AUC0-4)
Time Frame: 0 to 4 hours post-dose
Population: Some participants data was not included in the analysis due to having too few/insufficient data
Measure: Mean (Standard Deviation); unit: degree Celsius*Time
Arm/Group | Ibuprofen | Acetaminophen
Number analyzed (Participants) | 44 | 42
degree Celsius*Time | -4.4 (2.59) | -2.6 (2.02)

6. Secondary Outcome: Time to Afebrility (in Hours)
Description: Tme to afebrility (temperature less than 100.4 ºF [38 ºC]) in patients receiving intravenous ibuprofen and APAP.
Time Frame: 4 Hour post treatment
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Ibuprofen | Acetaminophen
Number analyzed (Participants) | 47 | 53
Hours | 2.2 (0.47) | 3.3 (0.67)

7. Secondary Outcome: Number of Afebrile and Febrile Subject at 4 Hours Post-Dose
Description: Number of Afebrile and Febrile Subject at 4 Hours Following Treatment
Time Frame: 4 Hours Post-Dose
Population: Some participants data was not included in the analysis due to having too few/insufficient data
Measure: Number; unit: participants
Arm/Group | Ibuprofen | Acetaminophen
Number analyzed (Participants) | 46 | 51
participants
  Afebrile Subjects at 4 hours | 43 | 40
  Febrile at 4 Hours | 3 | 11

ADVERSE EVENTS:
Arm/Group | Ibuprofen | Acetaminophen
Serious Adverse Events (participants affected / at risk) | 2/47 | 2/53
Other Adverse Events (participants affected / at risk) | 28/47 | 22/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibuprofen (N=47) | Acetaminophen (N=53)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Abdoimnal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Transaminases Increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibuprofen (N=47) | Acetaminophen (N=53)
Vomiting (Gastrointestinal disorders) | 3 (4) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 2 (2) | 2 (2)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 1 (1)
Blood Albumin Decreased (Investigations) | 2 (2) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 2 (2)
Oxygen Saturation Decreased (Investigations) | 2 (2) | 0 (0)
Infusion Site Pain (General disorders) | 5 (7) | 0 (0)
Hypokaelmia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No